CLINICAL TRIAL: NCT03692533
Title: Role of Immunohistochemical Markers , Geminin and Mcm2 in Prognosis of Renal Cell Carcinoma, and Its Clinicopathological Correlation. A Prospective Controlled Study
Brief Title: Role of Geminin and Mcm-2 in Prognosis of Renal Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelghany Allam, Assistant lecturer, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Geminin and Mcm-2 in RCC
Record Dates: First submitted 2018-09-20; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Renal Cell Carcinoma
Keywords: Geminin, prognosis
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Immunohistochemistry

STUDY DESIGN:
Intervention Model Description: 2 groups : Group A include cases and Group B includes controls
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group (A) [study cases] Adult patients who will undergo radical or partial nephrectomy.for primary renal cell carcinoma.
  Interventions: Diagnostic Test: Immunohistochemistry
- Group B (Active Comparator): Group (B) [control cases] Adult patients who will undergo simple nephrectomy for benign causes
  Interventions: Diagnostic Test: Immunohistochemistry

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry — Histopathological study and evaluation:
  For each case, the tissue samples will be evaluated by the pathologist for detecting the histopathology and in cases of malignant renal spicemens the pathologist will also assess the histologic type, Fuhrman nuclear grade, cellular invasion of perinephric fat, and the extent of any vascular invasion seen by microscopy.
  Immunohistochemistry:
  Immunohistochemical staining will be performed by using the following antibodies: Geminin and Minichromosome maintenance-2 (MCM-2).
  Evaluation of the immunohistochemical staining will be performed by light microscopy. The interpretation of immuno-reactivity will be performed in a quantitative manner by analyzing the extent of the staining positivity of the tumor cells. Immuno-staining of greater than 10% of tumor cells is required for scoring as a positive case.

SUMMARY:
The study aim is to prospectively assess the prognostic significance of immunohistochemical markers Geminin and Mcm-2 in cases of renal cell carcinoma and to detect its clinicopathological correlation.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is one of the most common urological malignancies. Approximately 338,000 people are diagnosed with RCC worldwide each year, representing approximately 2-3 % of all cancers.

RCC can be classified into non-epithelial and epithelial, according to cell origin. The four major types are of epithelial origin includes: clear cell renal carcinoma (ccRCC), papillary, chromophobe renal carcinoma (chRCC) and collecting duct carcinoma. The most common subtype of RCC is ccRCC which accounts for approximately 70-80% of all renal cell carcinomas.

Prognostic factors for RCC can be classified into: anatomical, histological, clinical, and molecular factors. Anatomical factors include tumor size, venous invasion, renal capsular invasion, adrenal involvement, Lymph node and distant metastasis. Histological factors include tumour grade, RCC subtype, sarcomatoid features, microvascular invasion, tumour necrosis, and invasion of the collecting system. Clinical factors include performance status, local symptoms, cachexia, anaemia, platelet count, neutrophil/lymphocyte ratio, C-reactive protein (CRP) and serum albumin.

As regard the molecular factors, numerous markers such as carbonic anhydrase IX, vascular endothelial growth factor (VEGF), hypoxia-inducible factor (HIF), Ki67, PTEN (phosphatase and tensin homolog), osteopontin and other cell cycle and proliferative markers are being investigated.

The efficiency and accuracy of biomarkers studies using immunohistochemical and tissue microarray techniques are still variable and unclear in regards to prognostic significance in patients with renal tumors. Multiple biomarkers shown to be significant to assess diagnosis and prognosis in these patients and other were not significant.

In the RCC cell cycle, minichromosome maintenance 2 (Mcm2), Geminin define the proliferative state. Investigators are able to determine differential levels of expression of various markers in normal tissue compared with indolent and aggressive tumors. Among platforms used in determining the presence of biological markers in surgical pathology specimens, immunohistochemistry is perhaps the most commonly available tool in the routine diagnostic laboratory. Immunohistochemistry allows detection of antigens expressed on tumor cells, hence permitting characterization of the tumor.

This study was designed to assess the prognostic significance of Geminin and Mcm-2 in cases of renal cell carcinoma and to assess its clinicopathological correlation.

ELIGIBILITY:
Inclusion criteria:

* Adult patients who will undergo radical or partial nephrectomy for primary Renal cell carcinoma (Group A).
* Adult patients who will undergo simple nephrectomy for benign causes (Group B).

Exclusion criteria:

* Patients with secondary renal metastasis.
* Patients with metastatic spread at time of presentation or operation.
* Patients with renal urothelial carcinomas.
* Children with renal tumors (less than 18 years).
* Patients who are unfit for surgical treatment.
* Patients who are refusing surgical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants that develops recurrence of tumor as assessed by Multi slice CT | 2 years
  Number of patients that develops recurrent tumor after partial or radical nephrectomy as diagnosed by Multi slice CT will be assessed
Number of participants that develops Tumor metastasis as assessed by Multi slice CT | 2 years
  Number of patients that develops tumor metastasis after partial or radical nephrectomy as diagnosed by Multi slice CT will be assessed

REFERENCES:
- [Background] Motzer RJ, Escudier B, McDermott DF, George S, Hammers HJ, Srinivas S, Tykodi SS, Sosman JA, Procopio G, Plimack ER, Castellano D, Choueiri TK, Gurney H, Donskov F, Bono P, Wagstaff J, Gauler TC, Ueda T, Tomita Y, Schutz FA, Kollmannsberger C, Larkin J, Ravaud A, Simon JS, Xu LA, Waxman IM, Sharma P; CheckMate 025 Investigators. Nivolumab versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1803-13. doi: 10.1056/NEJMoa1510665. Epub 2015 Sep 25. PMID 26406148
- [Result] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Result] Humphrey PA, Moch H, Cubilla AL, Ulbright TM, Reuter VE. The 2016 WHO Classification of Tumours of the Urinary System and Male Genital Organs-Part B: Prostate and Bladder Tumours. Eur Urol. 2016 Jul;70(1):106-119. doi: 10.1016/j.eururo.2016.02.028. Epub 2016 Mar 17. PMID 26996659
- [Result] Ljungberg B, Cowan NC, Hanbury DC, Hora M, Kuczyk MA, Merseburger AS, Patard JJ, Mulders PF, Sinescu IC; European Association of Urology Guideline Group. EAU guidelines on renal cell carcinoma: the 2010 update. Eur Urol. 2010 Sep;58(3):398-406. doi: 10.1016/j.eururo.2010.06.032. Epub 2010 Jul 12. PMID 20633979
- [Result] Sun M, Shariat SF, Cheng C, Ficarra V, Murai M, Oudard S, Pantuck AJ, Zigeuner R, Karakiewicz PI. Prognostic factors and predictive models in renal cell carcinoma: a contemporary review. Eur Urol. 2011 Oct;60(4):644-61. doi: 10.1016/j.eururo.2011.06.041. Epub 2011 Jun 30. PMID 21741163
- [Result] Kim HL, Belldegrun AS, Freitas DG, Bui MH, Han KR, Dorey FJ, Figlin RA. Paraneoplastic signs and symptoms of renal cell carcinoma: implications for prognosis. J Urol. 2003 Nov;170(5):1742-6. doi: 10.1097/01.ju.0000092764.81308.6a. PMID 14532767
- [Result] Haas NB, Manola J, Uzzo RG, Flaherty KT, Wood CG, Kane C, Jewett M, Dutcher JP, Atkins MB, Pins M, Wilding G, Cella D, Wagner L, Matin S, Kuzel TM, Sexton WJ, Wong YN, Choueiri TK, Pili R, Puzanov I, Kohli M, Stadler W, Carducci M, Coomes R, DiPaola RS. Adjuvant sunitinib or sorafenib for high-risk, non-metastatic renal-cell carcinoma (ECOG-ACRIN E2805): a double-blind, placebo-controlled, randomised, phase 3 trial. Lancet. 2016 May 14;387(10032):2008-16. doi: 10.1016/S0140-6736(16)00559-6. Epub 2016 Mar 9. PMID 26969090
- [Result] Kim HL, Han KR, Zisman A, Figlin RA, Belldegrun AS. Cachexia-like symptoms predict a worse prognosis in localized t1 renal cell carcinoma. J Urol. 2004 May;171(5):1810-3. doi: 10.1097/01.ju.0000121440.82581.d3. PMID 15076282
- [Result] Sim SH, Messenger MP, Gregory WM, Wind TC, Vasudev NS, Cartledge J, Thompson D, Selby PJ, Banks RE. Prognostic utility of pre-operative circulating osteopontin, carbonic anhydrase IX and CRP in renal cell carcinoma. Br J Cancer. 2012 Sep 25;107(7):1131-7. doi: 10.1038/bjc.2012.360. Epub 2012 Aug 23. PMID 22918393
- [Result] Choueiri TK, Escudier B, Powles T, Tannir NM, Mainwaring PN, Rini BI, Hammers HJ, Donskov F, Roth BJ, Peltola K, Lee JL, Heng DYC, Schmidinger M, Agarwal N, Sternberg CN, McDermott DF, Aftab DT, Hessel C, Scheffold C, Schwab G, Hutson TE, Pal S, Motzer RJ; METEOR investigators. Cabozantinib versus everolimus in advanced renal cell carcinoma (METEOR): final results from a randomised, open-label, phase 3 trial. Lancet Oncol. 2016 Jul;17(7):917-927. doi: 10.1016/S1470-2045(16)30107-3. Epub 2016 Jun 5. PMID 27279544
- [Result] Wilkerson ML, Lin F, Liu H, Cheng L. The application of immunohistochemical biomarkers in urologic surgical pathology. Arch Pathol Lab Med. 2014 Dec;138(12):1643-65. doi: 10.5858/arpa.2014-0078-RA. PMID 25427043
- [Result] Dudderidge TJ, Stoeber K, Loddo M, Atkinson G, Fanshawe T, Griffiths DF, Williams GH. Mcm2, Geminin, and KI67 define proliferative state and are prognostic markers in renal cell carcinoma. Clin Cancer Res. 2005 Apr 1;11(7):2510-7. doi: 10.1158/1078-0432.CCR-04-1776. PMID 15814627
- [Result] Alexiev BA, Drachenberg CB. Clear cell papillary renal cell carcinoma: Incidence, morphological features, immunohistochemical profile, and biologic behavior: A single institution study. Pathol Res Pract. 2014 Apr;210(4):234-41. doi: 10.1016/j.prp.2013.12.009. Epub 2014 Jan 9. PMID 24485757